CLINICAL TRIAL: NCT02388269
Title: A Randomized, Single Centre, Double-blind, Parallel, Sham-controlled Pilot Study of the gammaCore®-G, a Non-invasive Vagus Nerve Stimulator Device for Treatment of Symptoms Caused by Functional Dyspepsia or Irritable Bowel Syndrome
Brief Title: A Randomized, Single Centre, Double-blind, Parallel, Sham-controlled Pilot Study Using gammaCore®-G
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ElectroCore INC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: GG-007
Record Dates: First submitted 2015-02-18; First posted 2015-03-13 (Estimated); Results first posted 2018-02-06 (Actual); Last update posted 2018-03-07 (Actual); Status verified 2018-02

CONDITIONS: Dyspepsia; Irritable Bowel Syndrome
MeSH Terms: conditions — Dyspepsia; Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- gammaCore®-G (Active Comparator): The user/operator applies the gammaCore®-G device to the skin on the right side and left side of the neck. The 2 stimulations should be performed on the same side of the neck before stimulating the other side. This is also applies with the doses increase in the open label phase. The user applies conductive gel to the stimulation surfaces to maintain an uninterrupted conductive path from the stimulation surfaces to the skin.
  The device is capable of delivering multiple patient treatments (doses). Each dose consists of 90 seconds of stimulation; for each dose, the device is active for 120 seconds before automatically stopping stimulation.The extra 30 seconds allows .
  Interventions: Device: gammaCore®-G
- gammaCore®-G sham (Sham Comparator): The sham device is a hand-held portable device that appears identical to the gammaCore®-G, in look, weight, visual and audible feedback, user application and control. It passes a low frequency (0.1 Hz) biphasic DC signal into the tissue, which can be felt as a tingling sensation but does not stimulate the vagus nerve or cause muscle contraction. Similar to the active device, the sensation becomes more pronounced as the amplitude is increased, until it is uncomfortable, at which point the amplitude is decreased slightly until tolerable.
  Like the active device, the sham device is a multi-use device capable programmed to deliver up to 150, 90-second "treatments" with a 30-second margin for set-up and operator adjustment of the "stimulation intensity".
  Interventions: Device: gammaCore®-G

INTERVENTIONS:
Device: gammaCore®-G — The gammaCore®-G device is a reusable, hand-held, portable device consisting of two 3.0 VDC batteries (not replaceable or user serviceable), signal generating and amplifying electronics, and two buttons for operator control of the signal amplitude. The device provides visible (light display) and audible feedback on device and stimulation status

SUMMARY:
A randomized, sham-controlled, single-centre pilot investigation designed to compare two parallel groups, gammaCore®-G (active treatment) and a sham, (inactive) treatment in subjects with FGIDs.

DETAILED DESCRIPTION:
This study, in subjects with FGIDs, is a , randomized, sham-controlled, single-centre pilot investigation designed to compare two parallel groups, gammaCore®-G (active treatment) and a sham, (inactive) treatment. The study period will begin with a two-week run-in period, followed by a four week comparative period when the subjects will randomized (1:1) to either active treatment or sham (inactive) treatment. The comparative period will be followed by an open label four week period, where the subjects in the sham treatment group will switch in treatment assignment to receive active treatment and the active group will continue to receive an active treatment.

ELIGIBILITY:
Inclusion Criteria:

The subjects have to meet all of the following criteria to be eligible to enter the investigation:

1. Signed Informed Consent Form
2. Age >18
3. Diagnose with FD or IB Rome III criteria
4. Is able to complete the diary, use the device and to follow study procedures
5. Dyspepsia inclusion criteria, functional dyspepsia according to Rome III Diagnostic Criteria for Functional Gastrointestinal Disorders, one or more of the following:

   * Bothersome postprandial fullness
   * Early satiation
   * Epigastric pain
   * Epigastric burning
   * No evidence of structural disease (including at upper endoscopy) that is likely to explain the symptoms * Criteria fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis
6. IBS inclusion criteria, Irritable Bowel Syndrome* according to Rome III Diagnostic Criteria for Functional Gastrointestinal Disorders
7. Recurrent abdominal pain or discomfort** at least 3 days/month in the previous 3 months associated with two or more of the following:

   * Improvement with defecation
   * Onset associated with a change in frequency of stool
   * Onset associated with a change in form (appearance) of stool
   * Criterion fulfilled for the last 3 months with symptom onset at least 6 months prior to diagnosis ** "Discomfort" means an uncomfortable sensation not described as pain.
8. In pathophysiology research and clinical trials, a pain/discomfort frequency of at least 2 days a week during screening evaluation is recommended for subject eligibility.

Exclusion Criteria:

Subjects meeting any of the following criteria will not be permitted to enter the investigation:

1. Any positive endoscopic findings such as abnormal biopsy findings and/or any other abnormal finding judged by the Investigator
2. Any positive findings after sigmoidoscopy or colonoscopy such as diverticulosis, inflammatory bowel disease or other abnormal finding judged by the Investigator.
3. Vagotomy at any location
4. Has a neck lesion (including lymphadenopathy), dysaesthesia, previous surgery or abnormal anatomy at the site gammaCore®-G treatment
5. Has known or suspected severe atherosclerotic cardiovascular disease, severe carotid artery disease (e.g. bruits or history of transient ischemic attack (TIA) or cerebral vascular accident CVA), congestive heart failure (CHF), known severe coronary artery disease or recent (5 years) myocardial infarction
6. Has an abnormal baseline ECG (e.g. second and third degree heart block, atrial fibrillation, atrial flutter, recent history of ventricular tachycardia or ventricular fibrillation, or clinically significant premature ventricular contraction
7. Has uncontrolled hypertension
8. Is currently implanted with an electrical and/or neurostimulator device, including but not limited to cardiac pacemaker or defibrillator, vagal neurostimulator, deep brain stimulator, spinal stimulator, bone growth stimulator, gastric stimulator or cochlear implant
9. Has a history of carotid endarterectomy or vascular neck surgery
10. Has been implanted with metal cervical spine hardware or has a metallic implant near the GammaCore®-G stimulation site
11. Has a recent (within 12 months) or repeated history of syncope
12. Has a recent (within 12 months) or repeated history of seizures
13. Has psychiatric or cognitive disorder and/or behavioural problems which in the opinion of the clinician may interfere with the study
14. Is pregnant, nursing, thinking of becoming pregnant during the study period
15. Is participating in any other therapeutic clinical investigation or has participated in a clinical trial within 30 days period prior to this study
16. Is a relative of or an employee of the investigator or the clinical study site
17. Used gammaCore®-G previously

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Owen Epstein, Prof., Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Free Hospital NHS Trust, Centre for Gastroenterology, 8th floor, Pond street, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- gammaCore®-G: Active Comparator: Active gammaCore device
  gammaCore active stimulation treatment
- gammaCore®-G Sham: Sham Comparator: sham gammaCore device
  gammaCore sham stimulation treatment
- Not Randomised: Subjects that were not randomised, i.e. screen failures
Period: Overall Study
Arm/Group | gammaCore®-G | gammaCore®-G Sham | Not Randomised
Started (Run-in period) | 41 | 40 | 10
Randomised Period | 41 | 40 | 0
Open Label | 37 | 38 | 0
Completed (completed = run-in + randomised + open label periods) | 32 | 38 | 0
Not Completed | 9 | 2 | 10
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — less than 50% stimulations | 1 | 0 | 0
Not completed — no diary data | 3 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0
Not completed — Screen Failure | 0 | 0 | 10

BASELINE CHARACTERISTICS:
Groups:
- gammaCore®-G Functional Dyspepsia; gammaCore®-G Irritable Bowel Syndrome: Active Comparator: Active gammaCore device
  gammaCore active stimulation treatment
- gammaCore®-G Sham Functional Dyspepsia; gammaCore®-G Sham Irritale Bowel Syndrome: Sham Comparator: sham gammaCore device
  gammaCore sham stimulation treatment
- Total: Total of all reporting groups
Arm/Group | gammaCore®-G Functional Dyspepsia | gammaCore®-G Sham Functional Dyspepsia | gammaCore®-G Irritable Bowel Syndrome | gammaCore®-G Sham Irritale Bowel Syndrome | Total
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.6 (14.39) | 33.9 (12.01) | 40.1 (13.78) | 41.1 (16.84) | 38.9 (14.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 16 | 15 | 56
  Male | 7 | 8 | 5 | 5 | 25
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white | 18 | 16 | 20 | 16 | 70
  black | 0 | 2 | 0 | 4 | 6
  asian | 2 | 1 | 1 | 0 | 4
  other | 0 | 1 | 0 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 20 | 20 | 21 | 20 | 81

OUTCOME MEASURES:

1. Primary Outcome: Symptom Changes in Subjects With Functional Gastrointestinal Disorder (Functional Dyspepsia and Irritable Bowel Syndrome)
Description: Global Overall Symptom (GOS) scale is self-reported. Patients grade overall severity of dyspepsia symptoms over a retrospective period of time. The scale uses a 7-point Likert scale ranging from minimum 1 = no problem to maximum 7 = very severe problem. Subjects assess how their stomach problems have been over the specific time period, and indicate severity of symptoms for 10 specific upper GI symptoms (epigastric pain, epigastric discomfort, heartburn, acid regurgitation, upper abdominal bloating, excessive belching, nausea, early satiety, postprandial fullness, other epigastric symptoms). Total minimum = 10 and total maximum = 70. The Irritable Bowel Syndrome Score (IBS) measures severity of symptoms by 5 questions: abdominal pain, number days with pain in every 10 days (multiplied by 10), abdominal distension, bowel movement satisfaction, interference with general life. Each question scores from 0 (not severe) to 100 (severe). Total score: Min = 0 healthy; Max = 500 severely sick.
Time Frame: Last 2 weeks in the 4 week Randomized period
Population: Intention To Treat population (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | gammaCore®-G | gammaCore®-G Sham
Number analyzed (Participants) | 37 | 39
units on a scale
  Functional Dyspepsia: number analyzed (Participants) | 18 | 20
  Functional Dyspepsia | -0.6 (0.62) | -1.29 (1.13)
  Irritable Bowel Syndrome: number analyzed (Participants) | 19 | 19
  Irritable Bowel Syndrome | -46.84 (89.91) | -40.24 (78.62)

2. Secondary Outcome: Quality of Life (QoL) Using the Functional Digestive Disorder Quality of Life (FDDQL)
Description: Compare Quality of Life in last 2 weeks in the randomized period with the run-in period, and compare of Quality of life in the open label period to randomization period using the Functional Digestive Disorder Quality of Life (FDDQL) questionnaire.
  The Functional Digestive Disorder Quality of Life (FDDQL) questionnaire is designed to measure Quality of Like (QOL) in patients with Functional Dyspepsia (FD) or Irritable Bowel Syndrome (IBS). The questionnaire is composed of 43 items (questions) investigating 8 dimensions: Daily activities, Anxiety, Diet, Sleep, Discomfort, Health, Coping and Stress. For the 43 items, patients rate the impact of their condition over the 8 dimensions from 1-5, where 1 = Not at all, 2 = A little Bit, 3 = Moderately, 4= Quite a bit, and 5 = Extremely. The mean score of the 8 dimensions is shown in the outcome measure data table.
Time Frame: Run-In (2 weeks), Randomized (4 weeks) and Open Label (4 weeks) period
Population: Intention To Treat population (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- gammaCore®-G FD; gammaCore®-G IBS: Active Comparator: Active gammaCore device
  gammaCore active stimulation treatment
- gammaCore®-G Sham FD; gammaCore®-G Sham IBS: Sham Comparator: sham gammaCore device
  gammaCore sham stimulation treatment
Arm/Group | gammaCore®-G FD | gammaCore®-G Sham FD | gammaCore®-G IBS | gammaCore®-G Sham IBS
Number analyzed (Participants) | 18 | 20 | 19 | 19
units on a scale
  Daily Activities Run-in | 3.1 (1.03) | 2.9 (0.83) | 2.9 (0.80) | 3.2 (0.90)
  Daily Activities - Randomized Period | 2.7 (1.06) | 2.4 (0.85) | 2.6 (0.84) | 2.7 (0.98)
  Daily Activities - Open label | 2.5 (1.01) | 2.0 (0.78) | 2.5 (1.10) | 2.4 (1.04)
  Anxiety - Run-in | 3.3 (0.92) | 3.3 (0.83) | 3.4 (0.94) | 3.2 (1.03)
  Anxiety - Randomized | 2.9 (0.88) | 2.9 (0.71) | 3.2 (1.04) | 3.0 (0.97)
  Anxiety - Open-label | 2.7 (0.97) | 2.7 (0.90) | 3.1 (1.13) | 2.6 (0.92)
  Diet - Run-in | 3.6 (1.05) | 3.8 (0.8) | 3.9 (0.98) | 3.7 (0.6)
  Diet - Randomized | 3.6 (0.99) | 3.3 (0.95) | 3.6 (1.02) | 3.6 (0.70)
  Diet - Open-label | 3.4 (1.05) | 3.4 (1.07) | 3.3 (1.12) | 3.2 (0.82)
  Sleep - Run-in | 2.6 (0.96) | 2.7 (0.67) | 2.6 (0.88) | 2.8 (0.84)
  Sleep - Randomized | 2.5 (0.82) | 2.3 (1.05) | 2.4 (0.76) | 2.5 (0.76)
  Sleep - Open label | 2.3 (0.90) | 2.4 (1.02) | 2.4 (0.89) | 2.3 (0.95)
  Discomfort - Run-in | 3.5 (0.82) | 3.4 (0.72) | 3.7 (0.61) | 3.5 (0.74)
  Discomfort - Randomized | 3.4 (0.85) | 3.0 (0.59) | 3.2 (0.96) | 3.4 (0.69)
  Discomfort - Open label | 3.0 (0.83) | 2.9 (0.62) | 3.1 (1.09) | 2.8 (0.86)
  Health - Run-in | 2.8 (0.71) | 2.9 (0.63) | 2.6 (0.54) | 2.7 (0.72)
  Health - Randomized | 2.9 (0.91) | 3.1 (0.76) | 2.7 (0.71) | 2.8 (0.79)
  Health - Open label | 2.9 (0.87) | 3.0 (0.81) | 2.9 (0.82) | 2.9 (0.86)
  Coping - Run-in | 3.2 (0.85) | 3.5 (0.75) | 3.5 (0.91) | 3.5 (0.92)
  Coping - Randomized | 3.4 (0.91) | 3.1 (0.77) | 3.2 (1.04) | 3.4 (0.82)
  Coping - Open label | 3.0 (0.89) | 3.0 (0.81) | 3.3 (1.20) | 3.1 (0.97)
  Stress - Run-in | 3.5 (0.83) | 3.5 (1.05) | 3.3 (1.16) | 3.1 (1.03)
  Stress - Randomized | 3.5 (0.72) | 3.6 (1.07) | 3.2 (1.05) | 3.2 (1.05)
  Stress - Open label | 3.6 (0.90) | 3.4 (0.99) | 3.2 (1.15) | 3.1 (1.01)

3. Secondary Outcome: Change in Frequency of Symptoms Using the Short-Form Leeds Dyspepsia Questionnaire (SFLDQ)
Description: Compare last 2 weeks in randomized period with the run-in period; & compare open label period to randomization period using Short-Form Dyspepsia Questionnaire (SFLDQ).The SFLDQ is a validated, self-completed questionnaire that measures frequency and severity of dyspepsia. The questionnaire comprises of 5 questions, questions 1 to 4 are about the patients dyspeptic symptoms and question 5 is about the most troublesome symptom for the patient. Questions 1 to 4 comprise of two stems concerning 'frequency' (how often the subject has the symptom over the last 2 months) and 'severity' (how often has this symptom interfered with normal activities over the last 2 months). Subjects choose from: Not at all, less than monthly, between monthly & weekly, between weekly & daily, more than daily or no response. In question 5 the subject reports which symptoms has been most troublesome for each of the study periods. Results for Question 5 of the SFLDQ are reported separately in outcome measure 7.
Time Frame: Run-In (2 weeks), Randomized (4 weeks) and Open Label (4 weeks) period
Population: Intention to Treat
Measure: Count of Participants; unit: Participants
Groups:
- Frequency of Symptoms Over Last 2 Months - ACTIVE: Active Comparator: Active gammaCore device How often have you had this symptom over the last 2 months?
- Frequency of Symptoms Over the Last 2 Months - SHAM: Sham Comparator: sham gammaCore device How often have you had this symptom over the last 2 months?
- Interference With Normal Activities - ACTIVE: Active Comparator: Active gammaCore device How often has this symptom interfered with your normal activities over the last 2 months?
- Interference With Normal Activities - SHAM: Sham Comparator: sham gammaCore device How often has this symptom interfered with your normal activities over the last 2 months?
Arm/Group | Frequency of Symptoms Over Last 2 Months - ACTIVE | Frequency of Symptoms Over the Last 2 Months - SHAM | Interference With Normal Activities - ACTIVE | Interference With Normal Activities - SHAM
Number analyzed (Participants) | 18 | 20 | 18 | 20
Participants
  INDIGESTION:Run-in - Not at all | 1 | 0 | 2 | 3
  INDIGESTION:Run-in - Less than monthly | 0 | 1 | 2 | 1
  INDIGESTION:Run-in - Between weekly & monthly | 2 | 4 | 4 | 6
  INDIGESTION:Run-in -Between weekly & daily | 5 | 8 | 2 | 5
  INDIGESTION:Run-in - More than daily | 10 | 7 | 8 | 5
  INDIGESTION:Run-in - No response | 0 | 0 | 0 | 0
  INDIGESTION:Randomized- Not at all | 1 | 3 | 5 | 3
  INDIGESTION:Randomized- Less than monthly | 0 | 1 | 3 | 4
  INDIGESTION:Randomized- Between weekly & monthly | 1 | 1 | 0 | 5
  INDIGESTION:Randomized- Between weekly & daily | 11 | 8 | 5 | 3
  INDIGESTION:Randomized- More than daily | 3 | 6 | 3 | 4
  INDIGESTION:Randomized- No response | 2 | 1 | 2 | 1
  INDIGESTION:Open-label- Not at all | 1 | 3 | 5 | 5
  INDIGESTION:Open-label- Less than monthly | 2 | 2 | 2 | 3
  INDIGESTION:Open-label- Between monthly & weekly | 3 | 2 | 1 | 6
  INDIGESTION:Open-label- Between weekly an daily | 5 | 8 | 1 | 1
  INDIGESTION:Open-label- More than daily | 5 | 2 | 5 | 2
  INDIGESTION:Open-label- No response | 2 | 3 | 4 | 3
  HEARTBURN:Run-in- Not at all | 2 | 5 | 7 | 8
  HEARTBURN:Run-in- Less than monthly | 4 | 3 | 3 | 3
  HEARTBURN:Run-in- Between monthly & weekly | 6 | 3 | 2 | 2
  HEARTBURN:Run-in- Between weekly & daily | 5 | 6 | 4 | 5
  HEARTBURN:Run-in- More than daily | 1 | 3 | 2 | 1
  HEARTBURN:Run-in- No response | 0 | 0 | 0 | 1
  HEARTBURN:Randomised- Not at all | 6 | 5 | 11 | 10
  HEARTBURN:Randomised- Less than monthly | 6 | 5 | 4 | 1
  HEARTBURN:Randomised- Between monthly and weekly | 2 | 2 | 0 | 4
  HEARTBURN:Randomised- Between weekly and daily | 1 | 6 | 0 | 4
  HEARTBURN:Randomised- More than daily | 1 | 1 | 1 | 0
  HEARTBURN:Randomised- No response | 2 | 1 | 2 | 1
  HEARTBURN:Open-label- Not at all | 3 | 6 | 8 | 9
  HEARTBURN:Open-label- Less than monthly | 6 | 2 | 3 | 3
  HEARTBURN:Open-label- Between monthly & weekly | 2 | 4 | 0 | 4
  HEARTBURN:Open-label- Between weekly and daily | 4 | 5 | 2 | 1
  HEARTBURN:Open-label- More than daily | 1 | 0 | 1 | 0
  HEARTBURN:Open-label- No reposnse | 2 | 3 | 4 | 3
  REGURGITATION:Run-in- Not at all | 1 | 5 | 5 | 9
  REGURGITATION:Run-in- Less than monthly | 3 | 2 | 3 | 1
  REGURGITATION:Run-in- Between monthly and weekly | 7 | 4 | 5 | 2
  REGURGITATION:Run-in- Between weekly & daily | 5 | 3 | 3 | 6
  REGURGITATION:Run-in- More than daily | 2 | 6 | 2 | 2
  REGURGITATION:Run-in- No response | 0 | 0 | 0 | 0
  REGURGITATION:Randomized- Not at all | 3 | 5 | 7 | 7
  REGURGITATION:Randomized- Less than monthly | 4 | 4 | 3 | 5
  REGURGITATION:Randomized- Between monthly & weekly | 2 | 7 | 1 | 3
  REGURGITATION:Randomized- Between weekly & daily | 2 | 1 | 1 | 3
  REGURGITATION:Randomized- More than daily | 5 | 2 | 4 | 1
  REGURGITATION:Randomized- No response | 2 | 1 | 2 | 1
  REGURGITATION:Open-label- Not at all | 2 | 3 | 5 | 7
  REGURGITATION:Open-label- Less than monthly | 4 | 3 | 2 | 4
  REGURGITATION:Open-label- Between monthly & weekly | 2 | 4 | 3 | 4
  REGURGITATION:Open-label- Between weekly & daily | 4 | 6 | 3 | 1
  REGURGITATION:Open-label- More than daily | 4 | 1 | 1 | 1
  REGURGITATION:Open-label- No response | 2 | 3 | 4 | 3
  NAUSEA:Run-in- Not at all | 3 | 3 | 6 | 3
  NAUSEA:Run-in- Less than monthly | 1 | 0 | 2 | 1
  NAUSEA:Run-in- Between monthly & weekly | 2 | 3 | 2 | 4
  NAUSEA:Run-in- Bewteen weekly & daily | 5 | 7 | 3 | 8
  NAUSEA:Run-in- More than daily | 7 | 7 | 5 | 4
  NAUSEA:Run-in- No response | 0 | 0 | 0 | 0
  NAUSEA:Randomized- Not at all | 0 | 3 | 3 | 4
  NAUSEA:Randomized- Less than monthly | 3 | 3 | 4 | 5
  NAUSEA:Randomized- etween monthly & weekly | 3 | 5 | 2 | 3
  NAUSEA:Randomized- Between weekly & daily | 2 | 3 | 3 | 3
  NAUSEA:Randomized- More than daily | 8 | 5 | 4 | 4
  NAUSEA:Randomized- No response | 2 | 1 | 2 | 1
  Nausea: Open-label- Not at all | 0 | 1 | 5 | 4
  Nausea: Open-label- Less than monthly | 4 | 4 | 3 | 3
  Nausea: Open-label- Between monthly & weekly | 2 | 4 | 3 | 4
  Nausea: Open-label- Between weekly & daily | 7 | 6 | 2 | 5
  Nausea: Open-label- More than daily | 3 | 2 | 1 | 1
  Nausea: Open-label- No response | 2 | 3 | 4 | 3

4. Secondary Outcome: Use of Concomitant Medication (Intake and Dose) During the Course of the Study
Description: Compare last 2 weeks in randomised period with the run-in period, comparison open label period to randomization period. Concomitant medications were recorded and the number of subjects taking one or more concomitant medications is compared in the active and shams groups for both Functional Dyspepsia and Irritable Bowel Syndrome cohorts during the run-in, randomized and open label periods.
Time Frame: Run-In (2 weeks) and Randomized (4 weeks)
Population: Intent-to-Treat
Measure: Count of Participants; unit: Participants
Arm/Group | gammaCore®-G FD | gammaCore®-G Sham FD | gammaCore®-G IBS | gammaCore®-G Sham IBS
Number analyzed (Participants) | 20 | 20 | 21 | 20
Participants
  Subjects taking multiple medications in run-in | 15 | 18 | 18 | 18
  Subjects taking multiple medications in randomised | 17 | 17 | 19 | 17

5. Secondary Outcome: Symptom Change at 8 Weeks Compared to 4 Weeks (GOS Dyspepsia or IBS Severity Scoring System)
Description: as for outcome 1
Time Frame: Run-In (2 weeks), Randomized (4 weeks) and Open Label (4 weeks) period
Population: Intention To Treat (ITT)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | gammaCore®-G | gammaCore®-G Sham
Number analyzed (Participants) | 37 | 39
units on a scale
  Functional Dyspepsia: number analyzed (Participants) | 16 | 17
  Functional Dyspepsia | -0.03 (0.99) | -0.13 (0.66)
  Irritable Bowel Syndrome: number analyzed (Participants) | 16 | 18
  Irritable Bowel Syndrome | 0.27 (91.16) | -34.90 (65.84)

6. Secondary Outcome: Number of Participants With Adverse Events
Description: Summary of Treatment Emergent Adverse Events. Subjects were monitored for occurrence of adverse events from the start of the run-in period to the end of the open label period..
Time Frame: Run-In (2 weeks), Randomized (4 weeks) and Open Label (4 weeks) period
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Functional Dyspepsia Cohort Active: Functional Dyspepsia Cohort - Active gammacore
- Functional Dyspepsia Cohort Sham: Functional Dyspepsia Cohort - Sham gammacore
- Irritable Bowel Syndrome Cohort: Irritable Bowel Syndrome Cohort - Active gammacore
- Irritable Bowel Syndrome Cohort Sham: Irritable Bowel Syndrome Cohort - Sham gammacore
- Total Active Gammacore: Total Active gammacore - Functional Dyspepsia + Irritable Bowel Syndrome
- Total Sham Gammacore: Total Sham gammacore - Functional Dyspepsia + Irritable Bowel Syndrome
Arm/Group | Functional Dyspepsia Cohort Active | Functional Dyspepsia Cohort Sham | Irritable Bowel Syndrome Cohort | Irritable Bowel Syndrome Cohort Sham | Total Active Gammacore | Total Sham Gammacore
Number analyzed (Participants) | 20 | 20 | 21 | 20 | 41 | 40
Participants
  At least one event | 15 | 13 | 16 | 16 | 31 | 29
  At least one related event | 10 | 10 | 14 | 10 | 24 | 20
  At least one adverse device effect | 10 | 10 | 14 | 10 | 24 | 20
  At least one severe event | 4 | 2 | 7 | 2 | 11 | 4
  At least one serious event | 0 | 0 | 0 | 0 | 0 | 0
  At least one event leading to discontinuation | 3 | 0 | 3 | 1 | 6 | 1

7. Secondary Outcome: Change in Frequency of Symptoms Using the Short-Form Leeds Dyspepsia Questionnaire (SFLDQ)
Description: Short-Form Leeds Dyspepsia Questionnaire (SFLDQ): Question 5: Most Troublesome Symptom.
  In question five of the SFLDQ the subject reports which of the symptoms has been most troublesome to them, this is also reported for each of the study periods. (Note: results of questions 1-4 of the SFLDQ are reported separately in outcome measure 3.)
Time Frame: Run-In (2 weeks), Randomized (4 weeks) and Open Label (4 weeks) period
Measure: Count of Participants; unit: Participants
Groups:
- gammaCore®-G: Active Comparator: Active gammaCore device
  gammaCore active stimulation treatment - Functional Dyspepsia Cohort
- gammaCore®-G Sham: Sham Comparator: sham gammaCore device
  gammaCore sham stimulation treatment - Functional Dyspepsia Cohort
Arm/Group | gammaCore®-G | gammaCore®-G Sham
Number analyzed (Participants) | 18 | 20
Participants
  Run-in - Indigestion | 8 | 6
  Run-in - Heartburn | 1 | 1
  Run-in - Regurgitation | 1 | 2
  Run-in - Nausea | 8 | 9
  Run-in - None of these have troubled me | 0 | 1
  Run-in Missing | 0 | 1
  Randomized - Indigestion | 4 | 6
  Randomized - Heartburn | 0 | 2
  Randomized - Regurgitation | 3 | 1
  Randomized - Nausea | 9 | 7
  Randomized - None of these have troubled me | 0 | 0
  Randomized - Missing | 2 | 4
  Open-Label - Indigestion | 7 | 7
  Open-Label - Heartburn | 0 | 2
  Open-Label - Regurgitation | 2 | 1
  Open-Label - Nausea | 6 | 7
  Open-Label - None of these have troubled me | 1 | 0
  Open-Label - Missing | 2 | 3

ADVERSE EVENTS:
Time Frame: Adverse Event data was captured from the data of signature of informed consent (day -14) until final study visit (day 56), a total of 10 weeks. Any AE that was when the subject completed the study or was withdrawn from the study was followed-up until the AE was resolved or the clinical investigator decided that the AE was stable and needed no further follow up.
Arm/Group | gammaCore®-G FD | gammaCore®-G Sham FD | gammaCore®-G IBS | gammaCore®-G Sham IBS
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/21 | 0/20
Other Adverse Events (participants affected / at risk) | 15/20 | 13/20 | 16/21 | 16/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | gammaCore®-G FD (N=20) | gammaCore®-G Sham FD (N=20) | gammaCore®-G IBS (N=21) | gammaCore®-G Sham IBS (N=20)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blepharospasm (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis Allergic (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mydriasis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain Upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Food Poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritable bowel syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Odynophagia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Paraethesia Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tenderness (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Stress Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
MuscleTwitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Pain in Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 5 (5) | 2 (2) | 2 (2)
Headache (Nervous system disorders) | 5 (5) | 4 (4) | 5 (5) | 5 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Hypokinesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Panic Attack (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Respiratory Tract Ulceration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eczema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Skin Irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 3 (3) | 4 (4)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less